CLINICAL TRIAL: NCT00809341
Title: Treatment Intensification With R-ICE and High-Dose Cyclophosphamide for Diffuse Large B-Cell Non-Hodgkin's Lymphoma Based on Early [18F] FDG-PET Scanning
Brief Title: R-ICE and High-Dose Cyclophosphamide With PET/CT for Diffuse Large B-Cell Non-Hodgkin's Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: J0802; NA_00013656 (Other: JHMIRB); J0802 (Other: SKCCCRO)
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Results first posted 2018-09-25 (Actual); Last update posted 2018-09-25 (Actual); Status verified 2018-09

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: B-Cell; non-Hodgkin's; Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma | interventions — Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; Ifosfamide; Carboplatin; Etoposide; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PET Negative (Active Comparator): R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone) or an equivalent anthracycline-containing regimen for 3 cycles, followed by PET scan. Participants with a negative PET scan will complete their chemotherapy regimen as prescribed by their oncologist.
  Interventions: Biological: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Procedure: PET scan
- PET Positive (Active Comparator): R-CHOP (rituximab, cyclophosphamide, doxorubicin, vincristine, prednisone) or an equivalent anthracycline-containing regimen for 3 cycles, followed by PET scan. Participants with a positive PET scan will receive two cycles of R-ICE (rituximab, ifosfamide, carboplatin, etoposide) followed by HiCy (high-dose cyclophosphamide).
  Interventions: Biological: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone; Drug: Ifosfamide; Drug: Carboplatin; Drug: Etoposide; Drug: High-dose cyclophosphamide; Procedure: PET scan

INTERVENTIONS:
Biological: Rituximab — 375 mg/m^2 on Day 1 of each cycle as part of R-CHOP or R-ICE. Also given 375 mg/m^2 on Days 1, 30, and 37 as part of HiCy.
  Other Names: Rituxan
Drug: Cyclophosphamide — 750 mg/m^2 on Day 1 of each cycle as part of R-CHOP.
  Other Names: Cytoxan
Drug: Doxorubicin — 50 mg/m^2 on Day 1 of each cycle as part of R-CHOP.
  Other Names: Adriamycin; Hydroxydaunorubicin
Drug: Vincristine — 1.4 mg/m^2 on Day 1 of each cycle as part of R-CHOP.
  Other Names: Oncovin
Drug: Prednisone — 100 mg/day on Days 1-5 of each cycle as part of R-CHOP.
Drug: Ifosfamide — 2000 mg/m^2/day on Days 1-3 of each cycle as part of R-CHOP.
  Other Names: Ifex
  Arms: PET Positive
Drug: Carboplatin — Given on Day 2 of each cycle as part of R-CHOP. Dosed according to renal function.
  Other Names: Paraplatin
  Arms: PET Positive
Drug: Etoposide — 100 mg/m^2/day on Days 1-3 of each cycle as part of R-CHOP.
  Other Names: VP-16
  Arms: PET Positive
Drug: High-dose cyclophosphamide — 50 mg/kg/day on Days 2-5 of HiCy.
  Other Names: HiCy
  Arms: PET Positive
Procedure: PET scan — Performed once between Days 16-20 of cycle 3 of R-CHOP.
  Other Names: FDG-PET

SUMMARY:
This research is being done to see if a PET scan that is obtained after 3 cycles of a standard chemotherapy regimen can help guide treatment for patients with a blood disease called Non-Hodgkin's Lymphoma.

The standard treatment for newly diagnosed lymphoma is 6 to 8 cycles of chemotherapy like the CHOP combination (Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone). This regimen can cure about half of patients with lymphoma, but in many others disease relapses (comes back). Relapses are generally treated with more chemotherapy.

We believe that a PET scan (a type of imaging study that "lights up" in areas of cells with high activity such as lymphoma), may identify patients early who are at high risk of relapse.

The purpose of this research study is to find out if people whose treatment is changed early to an intensification regimen (high dose chemotherapy) based on a positive PET scan will have longer remissions than they would if they did not receive that high dose chemotherapy.

DETAILED DESCRIPTION:
Patients will receive 3 cycles of chemotherapy prior to mid-treatment PET-CT. Rituximab-CHOP, or an equivalent regimen must be used. During the third cycle of Rituximab-CHOP chemotherapy, a PET-CT scan will be performed. The PET scan will be designated as negative or positive. Based on the results, patients will either complete standard dose therapy or receive two cycles of R-ICE followed by high dose cyclophosphamide and rituximab.

A repeat PET-CT is required between 4 to 6 weeks following treatment completion. Patients will be followed-up every 4 months for 2 years, then every 6 months for one year, then annually until 5 years.

ELIGIBILITY:
Inclusion Criteria:

* One of the following Biopsy-confirmed, aggressive non-Hodgkin's lymphoma

  1. Diffuse large B-cell lymphoma
  2. Mediastinal (thymic) B-cell lymphoma
* Any stage (I through IV) as defined by the Ann Arbor staging system
* ECOG performance status of 0 to 2
* Radiographically measurable disease
* No more than 3 cycles of chemotherapy for lymphoma
* Greater than or equal to 18 years
* Adequate pulmonary, cardiac, hepatic, or renal function
* HIV antibody negative
* Women- Not pregnant or breastfeeding
* Men of reproductive potential must agree to use contraception

Exclusion Criteria:

* Patients with the following aggressive lymphomas are not eligible:

  1. Mantle cell
  2. Lymphoblastic
  3. Burkitt's
  4. Mycosis fungoides/Sezary's syndrome
  5. HTLV-1 associated T-cell leukemia/lymphoma
  6. Primary CNS lymphoma
  7. HIV-associated lymphoma
  8. Transformed lymphomas
  9. Immunodeficiency-associated lymphomas
* Previous diagnosis of another hematologic malignancies
* Progressive disease on CHOP or Rituximab-CHOP
* Active CNS involvement by lymphoma
* Serious co-morbid disease that could preclude full participation in study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lode Swinnen, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant was deemed ineligible and therefore not assigned to intervention. One participant withdrew informed consent prior to starting the study.
Groups:
- PET Negative; PET Positive: Patients with newly diagnosed diffuse large B-cell non-Hodgkin's lymphoma that have received 3 cycles of R-CHOP, or an equivalent anthracycline-containing regimen (e.g. R-CHOEP, R-EPOCH), will have a whole-body PET-CT scan performed to determine PET-positive or PET-negative status. These patients will then be assigned to a treatment arm based on the PET-positive or PET-negative status.
Period: Overall Study
Arm/Group | PET Negative | PET Positive
Started | 20 | 5
Completed | 20 | 4
Not Completed | 0 | 1
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PET Negative | PET Positive | Total
Number analyzed (Participants) | 20 | 5 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 4 | 19
  >=65 years | 5 | 1 | 6
Age, Continuous [Median (Full Range); unit: years] | 52.5 [23 to 72] | 50 [26 to 66] | 52 [23 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 | 9
  Male | 12 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival in Patient Receiving Early Treatment Intensification Based on a Positive Mid-treatment PET Scan
Time Frame: 2 years
Population: The study was placed on hold to determine a quantitative method for the evaluation of PET scan results. No decision was reached on the evaluation mechanism for the PET scans, so the study was terminated. Data for this outcome was not collected because a standardized evaluation mechanism for the PET scans was not found.
Arm/Group | PET Negative | PET Positive
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Overall Survival in Patients Whose Treatment is Determined on the Basis of a Mid-treatment [18F] FDG-PET Scan Result.
Time Frame: 5 years
Population: as for outcome 1
Arm/Group | PET Negative | PET Positive
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years
Arm/Group | PET Negative | PET Positive
All-Cause Mortality (participants affected / at risk) | 1/20 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/20 | 3/5
Other Adverse Events (participants affected / at risk) | 0/20 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PET Negative (N=20) | PET Positive (N=5)
Febrile Neutropenia (Infections and infestations) | 0 (0) | 2 (2)
Hemorrhage, CNS (Nervous system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes